CLINICAL TRIAL: NCT01638832
Title: Association of Non-alcoholic Fatty Liver Disease and Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JWGUHMED1-005
Record Dates: First submitted 2012-07-05; First posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: NASH; coronary artery disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transient Elastography (FibroScan), Echosens, Paris, France
Device: Controlled Attenuation Parameter (CAP), Echosens, Paris, France

SUMMARY:
This study will evaluate the association of non-alcoholic fatty liver disease and coronary artery disease. All patients presenting for coronary angiogram will receive the following examination:

* Transient Elastography and Controlled Attenuation Parameter using the FibroScan
* blood examination including biochemical markers The results of non-invasive liver steatosis and fibrosis measurement are compared with the results of coronary angiogram concerning the presence or absence of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years and older
* Written consent
* Coronary angiogram planned

Exclusion Criteria:

* Patients with mental diseases
* Pregnancy or lactation
* Ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Liver fibrosis scores I-IV (METAVIR)
  METAVIR fibrosis scores:
  I = mild fibrosis II = significant fibrosis III = advanced fibrosis IV = cirrhosis

SECONDARY OUTCOMES:
Steatosis fibrosis scores I-III
  Steatosis scores:
  0 = <5% I = 5-33% II = 33-66% III = >66%

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, MD, Principal Investigator — Klinikum der J. W. Goethe-Universität Frankfurt am Main
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Germany